CLINICAL TRIAL: NCT06782620
Title: Association Between Surgical Aortic Valve Replacement and Long-term Outcomes in 50 to 65-year-olds: Results of the AUTHEARTVISIT Study
Brief Title: Association Between Surgical Aortic Valve Replacement and Long-term Outcomes in 50 to 65-year-olds
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Alissa Florian, Dr. Alissa Florian, Medical University of Vienna
Other Study IDs: GS1-EK-4/722-2021
Record Dates: First submitted 2025-01-13; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Aortic Valve Replacement
Keywords: aortic valve replacement; mechanical AVR; biological AVR

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- sB-AVR: Patients with biological Aortic valve replacement
- sM-AVR: Patients with mechanical Aortic valve replacement

SUMMARY:
The goal of this observational study o is to compare outcomes after either biological or mechanical aortic valve replacement. The main question it aims to answer:

Is survival better after mechanical aortic valve replacement compared to biological aortic valve replacement? Are there less complications and reoperations after mechanical aortic valve replacement compared to biological aortic valve replacement? We perform a retrospective Data Collection of anonymized Austrian health insurance data.

DETAILED DESCRIPTION:
Objectives: In recent years, age recommendations for the utilization of biological prostheses rather than mechanical prostheses for surgical aortic valve replacement (sAVR) have been significantly reduced. This study evaluated survival rates, major adverse cardiac events (MACEs), and reoperation risks following surgical (sM-AVR) and biological (sB-AVR) AVR, with the aim of providing data to inform optimal prosthesis selection for middle-aged patients between 50 and 65 years.

Methods: A population-based cohort study was conducted using data from the Austrian Health System from 2010 to 2020. Patients undergoing isolated sAVR (n=3761) were categorized into sM-AVR (n=1018) and sB-AVR (n=2743) groups. Propensity score matching (PSM) was applied to balance covariates. The primary endpoint was all-cause mortality. The secondary endpoints included MACEs, reoperation, stroke, bleeding, and post-reoperation survival. Outcomes were assessed using Cox regression and Kaplan-Meier analyses.

ELIGIBILITY:
Inclusion Criteria:

* age between 50 and 65 years
* st. p. isolated biological or mechanical aortic valve replacement

Exclusion Criteria:

* transcatheter aortic valve implantation (TAVI; MEL codes DB025, DB026, DB021, or XN010) as index procedure
* age <50 or >65 years
* concomitant heart surgery or additional procedures during the index operation
* patients receiving a coronary artery stent (MEL codes DD050 or DD060) within four months before AVR

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * age between 50 and 65 years
  * st. p. isolated biological or mechanical aortic valve replacement
Sampling Method: Non-Probability Sample
Enrollment: 3761 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Survival | up to 12 years
  overall Survival

SECONDARY OUTCOMES:
reoperation-free survival | up to 12 years
  reoperation-free survival after either biological or mechanical AVR
reoperation | up to 12 years
  reoperation after either biological or mechanical AVR
MACEs | up to 12 years
  MACEs after either biological or mechanical AVR
heart failure | up to 12 years
  heart failure after either biological or mechanical AVR
embolic stroke or ICH | up to 12 years
  embolic stroke or ICH after either biological or mechanical AVR
myocardial infarction | up to 12 years
  myocardial infarction after either biological or mechanical AVR
non-embolic bleeding | up to 12 years
  non-embolic bleeding after either biological or mechanical AVR

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik J Ankersmit, Univ. Prof. Dr., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No